CLINICAL TRIAL: NCT02045628
Title: The Impact of an Investment Based Intervention on Weight-loss and Beliefs About Food in Patients Post Bariatric Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Surrey (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PB-PG-0212-27034
Record Dates: First submitted 2013-12-02; First posted 2014-01-27 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: Bariatric Surgery; Health Psychology
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investment intervention (Experimental): Those in the investment group will complete carefully framed questions designed to raise the salience of the investment they have made in their procedure at baseline and 3 months follow up. The content of this intervention will be tailored to the recent experiences of the patient (ie pre or post surgery).
  Interventions: Behavioral: Investment intervention
- Control (No Intervention): Those in the control group will receive usual care.

INTERVENTIONS:
Behavioral: Investment intervention — Those in the investment group will complete carefully framed questions designed to raise the salience of the investment they have made in their procedure at baseline and 3 months follow up. The content of this intervention will be tailored to the recent experiences of the patient (ie pre or post surgery).
  Arms: Investment intervention

SUMMARY:
Although obesity surgery is currently the most effective method for achieving weight loss, not all patients lose the desired amount of weight and some show weight regain. Previous pilot work by the lead researcher shows that successful weight loss is associated with the amount of investment the patient feels that they have made in their operation. For example, those who feel that it has taken more time and effort to organise, has cost more money, has been more disruptive to their family, social and work lives and has caused pain are more likely to lose weight after their operation. Therefore, it seems as if the greater the sense of investment, the greater the motivation to make the operation a success. The present study aims to build on these findings by encouraging weight loss surgery patients to focus on the investment they have made, thus making their investment more salient to them. Using a trial design, half the patients will be asked to rate and describe the investment they have made in their operation just before surgery (focusing on the time and effort to organise the surgery etc) and 3 months after surgery (focusing on time off work for recovery, disruption of family and friends, pain of surgery, pain of having the stitches removed etc). All patients will record their weight, beliefs about food, intentions to change their behaviour and actual eating and exercise behaviour at baseline then 3, 6 and 12 months follow up. The impact of the investment based intervention will then be assessed to explore whether focusing on the investment involved in having surgery improves patient health outcomes by one year.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or over
* having bariatric surgery at University College Hospital

Exclusion Criteria:

* if the patient does not understand English
* if the patient does not consent to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 12 months follow up.
  Excess weight loss at 12 months after bariatric surgery.

SECONDARY OUTCOMES:
Change in psychological outcomes | 12 month follow up
  Psychological issues relating to beliefs about food, intentions to change diet and exercise and actual diet and exercise behaviours.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Ogden, PhD, Principal Investigator — University of Surrey
Locations (1):
- University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hollywood A, Ogden J, Hashemi M. A randomised control trial assessing the impact of an investment based intervention on weight-loss, beliefs and behaviour after bariatric surgery: study protocol. BMC Obes. 2015 Mar 21;2:18. doi: 10.1186/s40608-015-0048-2. eCollection 2015. PMID 26217533